CLINICAL TRIAL: NCT06531967
Title: Development and Validation of a Prediction Model for Risk of Death in Kidney Transplant Recipients
Brief Title: Predicting Mortality in Kidney Transplant Recipients
Acronym: mBox
Status: Enrolling by invitation | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: mBox_001
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Death
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Necker hospital from Paris, France: Kidney recipients from Necker hospital
  Interventions: Other: No intervention
- Saint-Louis hospital from Paris, France: Kidney recipients from Saint-Louis hospital
  Interventions: Other: No intervention
- Bichat hospital from Paris, France: Kidney recipients from Bichat hospital
  Interventions: Other: No intervention
- Bretonneau hospital from Tours, France: Kidney recipients from Bretonneau hospital
  Interventions: Other: No intervention
- Toulouse hospital, France: Kidney recipients from Toulouse hospital
  Interventions: Other: No intervention
- KU Leuven, Belgium: Kidney recipients from KU Leuven
  Interventions: Other: No intervention
- Liege hospital from Belgium: Kidney recipients from Liege hospital
  Interventions: Other: No intervention
- Leiden University Medical Center from the Netherlands: Kidney recipients from Leiden University Medical Center
  Interventions: Other: No intervention
- Hospital of the University of Pennsylvania from Philadelphia, US: Kidney recipients from Hospital of the University of Pennsylvania
  Interventions: Other: No intervention
- Mayo Clinic from Phoenix, US: Kidney recipients from Mayo Clinic
  Interventions: Other: No intervention
- UCSF database: Kidney recipients data from real-world UCSF database
  Interventions: Other: No intervention
- AP-HP database: Kidney recipients data from real-world AP-HP database
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Accurately predicting kidney recipient risk of death has a crucial interest because of the organ shortage, the need to optimize allograft allocation by identifying high-risk patients who may not benefit from a transplant and improve the clinical decision-making after transplant to ensure that each patient survives as long as possible.

However, according to a literature review the investigators performed, studies attempting to develop a kidney recipient death prediction model suffer from many shortcomings, including the lack of key risk factors, use of biased registry data, small sample size, lack of external validation in different countries and subpopulations, and short follow-up.

The present study thus aimed to address these limitations and develop a robust, generalizable kidney recipient death prediction model.

DETAILED DESCRIPTION:
The number of individuals suffering from end-stage chronic renal disease (ESRD) worldwide has increased over time, exceeding seven million of patients in 2020. For individuals with ESRD, kidney transplantation is the best treatment in terms of patient survival, quality of life and from a cost-effective standpoint, as compared with dialysis, even in comorbid or elderly populations.

Although the number of kidney transplantations performed each year has increased as well, it follows a lower pace than the increase of individuals on the waiting-list, resulting in an organ shortage. There is therefore a need to optimize allograft allocation by identifying the high-risk patients who may not benefit from a transplant and improve the clinical decision-making after transplant to ensure that each patient survives as long as possible.

In this context, a kidney recipient death prediction model may improve transplant clinical practice, allowing for the ability to evaluate the individual risk of post transplant mortality, already before undergoing transplantation, thereby guiding decision making. However, developing such a model is a very difficult task, as death after kidney transplantation depends on many parameters, such as donor age, history or cause of death, imaging parameters, patients' past medical history (e.g. diabetes, dialysis duration, hypertension), patients' biological parameters, as well as the function of the allograft, which depends on patients' immunological factors, or allograft related parameters such as HLA mismatches or cold ischemia time.

The goal of the present study was therefore to identify the determinants of death after kidney transplantation, and to develop and validate a prediction model that would help optimize allograft allocation and post-transplant patient management, using a large, international, highly phenotyped cohort of kidney recipients with extensive data collection and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney recipients

Exclusion Criteria:

* Multi-organ transplantation
* Prior kidney transplant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, de novo, kidney recipients who received only a kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2004-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient death | Up to 10 years after kidney transplantation
  Patient death

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Principal Investigator — Paris Institute for Transplantation and Organ Regeneration (PITOR)
Locations (11):
- United States (3):
  - Department of Medicine, Mayo Clinic, Phoenix, Arizona
  - Bakar Computational Health Sciences Institute, University of California, San Francisco, California
  - Penn Transplant Institute, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Belgium (2):
  - Department of Nephrology and Renal Transplantation, University Hospitals Leuven, Leuven
  - Division of Nephrology, University Hospital Liège (CHU), Liège
- France (5):
  - Necker hospital, Paris
  - Saint-Louis hospital, Paris
  - Tenon hospital, Paris
  - Department of Nephrology and Organ Transplantation, Toulouse University Hospital, Toulouse
  - Department of Nephrology and Clinical Immunology, University Hospital of Tours, Tours
- Leiden Transplant Center, Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided